CLINICAL TRIAL: NCT00758719
Title: A Prospective Multicenter Lumbar Spine Fusion Study to Evaluate the Effectiveness of the Biomet Lumbar Spinal Fusion System
Brief Title: Evaluate Effectiveness of the Biomet Lumbar Spinal Fusion System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-045
Record Dates: First submitted 2008-09-09; First posted 2008-09-25 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Degenerative Disc Disease
Keywords: Spinal Fusion; Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Biomet Lumbar Spinal Fusion System in patients undergoing lumbar fusion surgery.

DETAILED DESCRIPTION:
All subjects enrolled in this study will receive the The Biomet Osteobiologic Treatment System which is comprised of the SpF® Spine Fusion Stimulator and any or all of the following can be utilized in the study: any Pedicle Screw System, autograft and an Interbody Spacer

ELIGIBILITY:
Inclusion Criteria:

1. The subject must, in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent.
2. The subject must be diagnosed with degenerative disc disease at up to 2 levels from L2-S1 inclusive and undergoing up to 2 level posterior lumbar spinal fusion surgery with or without anterior column fusion.
3. Subjects must be between 18 and 75 years of age.
4. The patient must be skeletally mature (epiphyses closed).

Exclusion Criteria:

1. Subject is pregnant, lactating or interested in becoming pregnant during the duration of the study.
2. Any active litigation.
3. Subject is currently involved in another investigational study.
4. Subject has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up.
5. Subject is incarcerated.
6. More than 2 prior spine surgeries/revision surgeries or any previous spinal fusions at levels being currently treated.
7. Traumatic instability.
8. Any parathyroid or metabolic bone disease.
9. Any active malignancy.
10. Osteopenia/Osteoporosis - All subjects will be screened for osteoporosis using SCORE (Simple Calculated Osteoporosis Risk Estimation) with a threshold value of 6. All subjects with a SCORE value greater than 6 will be referred for Dual-energy X-ray absorptiometry (DEXA) Scan. Subjects with a T-Score of £-1-2.5 will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is open to all patients with one or two level Degenerative Disease who are between the ages of 18 and 75.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Radiographic Fusion | 12 Month

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) change from baseline | 24 Months
  Mean VAS % change from baseline
Oswestry Disability Index change from baseline | 24 Month
  Oswestry Disability Index % change from baseline
Neurologic Assessment, Maintenance or improvement from baseline | 12 Month
Short Form Health Survey (SF-36) % change from baseline | 24 Month
Time to return to work | 24 month
Time to return to normal activity | 24 month
Narcotic Use | 24 month
  pre and post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Joel Batts, Study Director — Biomet Spine
Locations (4):
- United States (4):
  - Union Hospital Neurosurgical, Terre Haute, Indiana
  - Family Orthopedic Associates, Flint, Michigan
  - Orthopedics and Neurological Consultants, Inc, Columbus, Ohio
  - Neurological Associates of Waukesha, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided